CLINICAL TRIAL: NCT02134600
Title: OmegaChild - Omega-3 Supplementation to Children Now in Full Remission From a Previous Cancer; an Early Phase Dose-finding Study.
Brief Title: OmegaChild - Omega-3 Supplementation to Children Previously Treated for Cancer
Acronym: OmegaChild
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Per Kogner (Other)
Collaborators: Smartfish AS (Industry)
Responsible Party: Sponsor-Investigator, Per Kogner, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20130321
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pediatric Cancer
Keywords: Omega-3 fatty acids; DHA; EPA; Docosahexaenoic acid; Eicosapentaenoic acid; Childhood cancer; Body composition; Inflammation; Neuropsychiatric symptoms
MeSH Terms: conditions — Neoplasms; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega-3 enriched fruit juice (Experimental): Single arm study: Omega-3 enriched fruit juice in increasing dosage
  Interventions: Dietary Supplement: Omega-3 enriched fruit juice

INTERVENTIONS:
Dietary Supplement: Omega-3 enriched fruit juice — Different doses of omega-3 will be administered to five different groups:
  400, 800, 1200, 2400 and 3000 mg/m2.
  Other Names: Nutrifriend by Smartfish AS

SUMMARY:
The purpose of this study is to find an optimal dose of omega-3 that can be given to children who have completed cancer therapy. The future aim is to add omega-3 to conventional cancer treatment modalities and thereby hopefully increase the treatment efficacy, which will have to be addressed in subsequent phase-2 studies.

DETAILED DESCRIPTION:
The rationale for this phase-1 trial is to find an appropriate dose of omega-3 for future phase-2 studies. The investigators aim at defining a dose that can safely be given to children previously treated for cancer, and that does not cause unacceptable side effects. In a longer perspective, randomized control trials are planned where the supplement is given for longer periods of time, and in combination with conventional cancer treatment. In preparation for these trials, this dose finding study was designed that also evaluates compliance. Subsequently the investigators hope that this supplementation can be beneficial for children during both cancer treatment and after remission.

The study population consists of children judged to be in complete clinical remission from cancer. In a phase 1 trial, one usually uses healthy individuals as study subjects, but in pediatric studies this is not allowed. Therefore patients who are in full remission were chosen as study objects, but who still come to the clinic for regular follow-ups. This group of patients is relevant for this study since it represents all ages and base-line diets, all kinds of childhood cancers, and because they have suffered from cancer and in many cases still live with the severe consequences of it.

The study is designed to give five groups of eight individuals each different doses of omega-3 adjusted to body surface area. The first group starts out on a dose of omega-3 fatty acids that is similar to the generally recommended daily intake for adults (200-400 mg). A dose escalation is then done performed group wise. The highest possible dose in this study (2 x 3000mg/day at dose level 3000 mg/m2 to a child at 1.55 m2, 3871 mg/m2) is still lower than what has previously been given as maximum to children in other studies. The investigators will keep escalating the dose level within the study only as long as no unacceptable side effects are reported.

The administration is done orally by drinking 200 mL of omega-3 supplemented fruit juice daily. It has a good fruity taste, low amounts of sugar, and no fish flavour. This should facilitate treatment compliance for the children in particular compared to when omega-3 is given in capsules - the commonest choice in other studies, but less suitable for children. Compliance is important and not further jeopardized by trying to divide the fruit juice in less amounts than the whole package, but the individually prescribed dose as well as the actual amount ingested will be recorded and exact calculations used in the analysis of the study.

All study results are primarily evaluated on an intention-to-treat basis, but will also be calculated as treated per protocol and further calculated on the exact dose consumed over 90 days given the compliance in terms of consumed number of fruit juice packages.

ELIGIBILITY:
Inclusion Criteria:

1. 2-18 years old
2. Diagnosed with and now in complete clinical remission from any type of cancer
3. Completed conventional therapy according to specific protocols within three years
4. Spoken and written Swedish is understood by caregiver and/or child
5. Expected to attend clinical follow-ups the coming three months.
6. Performance Level: Karnofsky ≥ 60% for patients > 16 years of age and Lansky ≥ 60 for patients ≤16 years of age. Note: Neurologic deficits in patients with tumors of the CNS (central nervous system) must have been relatively stable for a minimum of 1 month prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
7. Written informed consent by all caregivers and if possible by the child after 7 years of age.

Exclusion Criteria:

1. Known coagulation disorder
2. Expected elective invasive surgery during the treatment
3. Allergic to: fish or fish oil, protein from cow milk, fruit juice from any of the included fruits (apple, pear, pomegranate, passion fruit, peach, aronia)
4. Supplementation of omega-3 during the last month
5. Regular intake of NSAIDs (nonsteroidal antiinflammatory drugs), aspirin (ASA) or vitamin D
6. Breastfeeding or pregnancy
7. Participates in other clinical trials where results may be altered by additional intervention

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09-02 (Actual)

PRIMARY OUTCOMES:
Omega-3 index | 3 months
  Omega-3 index is defined as % of DHA + EPA of total fatty acids in erythrocyte membranes.
  (DHA: Docosahexaenoic acid. EPA: Eicosapentaenoic acid).

SECONDARY OUTCOMES:
Adverse Events | 3 months
  Adverse events will be graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) v.4.

OTHER OUTCOMES:
Compliance | 3 months
  Compliance is calculated in percentage (%) using the number of fruit juice packages actually consumed (according to patient diary and interview) / number of packages prescribed (one or two daily pending dose level and body surface area).

CONTACTS AND LOCATIONS:
Overall Officials: Per Kogner, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Childhood Cancer Research Unit, Astrid Lindgren Children´s Hospital, Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Gleissman H, Segerstrom L, Hamberg M, Ponthan F, Lindskog M, Johnsen JI, Kogner P. Omega-3 fatty acid supplementation delays the progression of neuroblastoma in vivo. Int J Cancer. 2011 Apr 1;128(7):1703-11. doi: 10.1002/ijc.25473. Epub 2010 May 24. PMID 20499314
- [Background] Gleissman H, Johnsen JI, Kogner P. Omega-3 fatty acids in cancer, the protectors of good and the killers of evil? Exp Cell Res. 2010 May 1;316(8):1365-73. doi: 10.1016/j.yexcr.2010.02.039. Epub 2010 Mar 6. PMID 20211172
- [Background] Gleissman H, Yang R, Martinod K, Lindskog M, Serhan CN, Johnsen JI, Kogner P. Docosahexaenoic acid metabolome in neural tumors: identification of cytotoxic intermediates. FASEB J. 2010 Mar;24(3):906-15. doi: 10.1096/fj.09-137919. Epub 2009 Nov 4. PMID 19890019
- [Background] Lindskog M, Gleissman H, Ponthan F, Castro J, Kogner P, Johnsen JI. Neuroblastoma cell death in response to docosahexaenoic acid: sensitization to chemotherapy and arsenic-induced oxidative stress. Int J Cancer. 2006 May 15;118(10):2584-93. doi: 10.1002/ijc.21555. PMID 16353135